CLINICAL TRIAL: NCT01825447
Title: A Randomized, Single-Dose, Placebo-Controlled, Double-Blind, 3-Way Crossover Study to Determine the Relative Abuse Potential of Intravenous Oxycodone Hydrochloride Alone or in Combination With Intravenous Naltrexone Hydrochloride in Opioid Experienced Non-Dependent Subjects
Brief Title: A Study to Characterize the Abuse Liability of Intravenous Oxycodone Alone or in Combination With Intravenous Naltrexone in Healthy, Non-Dependent, Recreational Opioid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Lifetree Clinical Research Center, Salt Lake City, Utah (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B4981002
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: abuse potential; abuse liability; drug liking; oxycodone; naltrexone; intravenous; pharmacodynamic
MeSH Terms: interventions — Oxycodone; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment B (Experimental)
  Interventions: Drug: Oxycodone + Naltrexone
- Treatment C (Active Comparator)
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Placebo — 0.9% sodium chloride for injection x 1 dose administered intravenously (IV) push over 4 min.
  Arms: Treatment A
Drug: Oxycodone + Naltrexone — Oxycodone hydrochloride (HCl) 20 mg IV and naltrexone HCl 2.4 mg IV administered simultaneously x 1 dose IV push over 4 min.
  Arms: Treatment B
Drug: Oxycodone — Oxycodone HCl 20 mg for injection x 1 dose IV push over 4 min.
  Arms: Treatment C

SUMMARY:
The main purpose of this study is to simulate if oxycodone and naltrexone combination capsules (ALO-02) were to be tampered with by dissolving and then injecting intravenously for the purpose of getting high.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Non-dependent, recreational opioid users
* Must include at least one of these routes of administration: intranasal use on at least 3 occassions in the past year or intravenous use on at least 1 occasion in the past year before Screening (Visit 1).

Exclusion Criteria:

* Diagnosis of substance and/or alcohol dependence
* Subject has participated in, is currently participating in, or seeking treatment for substance and/or alcohol related disorder
* History of sleep apnea.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Drug Liking: Area Under Effect Curve (AUE) From 0-2 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100-point bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of
Drug Liking: Peak Effect (Emax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
High: Area Under Effect Curve (AUE) From 0-2 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
  High VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
High: Peak Effect (Emax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose

SECONDARY OUTCOMES:
Drug Liking: Area Under Effect Curve (AUE) From 0-1 Hour | 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100-point bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of
Drug Liking: Area Under Effect Curve (AUE) From 0-8 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
High: Area Under Effect Curve (AUE) From 0-1 Hour | pre-dose, 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  High VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
High: Area Under Effect Curve (AUE) From 0-8 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Take Drug Again: Peak Effect (Emax) | 12, 24 h post-dose
  Take Drug Again VAS is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100-point bipolar VAS with score ranging from 0 mm to 100 (score of 0 =
Take Drug Again: Mean Effect (Emean) | 12, 24 h post-dose
Overall Drug Liking: Peak Effect (Emax) | 12, 24 h post-dose
  Overall Drug Liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100-point VAS is used to assess response based on a score ranging from 0 to 100 (0 =
Overall Drug Liking: Mean Effect (Emean) | 12, 24 h post-dose
Any Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour | 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Any Drug Effects VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Any Drug Effects: Area Under Effect Curve (AUE) From 0-2 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h post-dose
Any Drug Effects: Area Under Effect Curve (AUE) From 0-8 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Good Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour | 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Good Drug Effects VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Good Drug Effects: Area Under Effect Curve (AUE) From 0-2 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h
Good Drug Effects: Area Under Effect Curve (AUE) From 0-8 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-1 Hour | 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Bad Drug Effects VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-2 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h
Bad Drug Effects: Area Under Effect Curve (AUE) From 0-8 Hours | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Feel Sick: Area Under Effect Curve (AUE) From 0-1 Hour | pre-dose, 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Feel Sick VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Feel Sick: Area Under Effect Curve (AUE) From 0-2 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h post-dose
Feel Sick: Area Under Effect Curve (AUE) From 0-8 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Nausea: Area Under Effect Curve (AUE) From 0-1 Hour | pre-dose, 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Nausea VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Nausea: Area Under Effect Curve (AUE) From 0-2 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h post-dose
Nausea: Area Under Effect Curve (AUE) From 0-8 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Sleepy: Area Under Effect Curve (AUE) From 0-1 Hour | pre-dose, 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Sleepy VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Sleepy: Area Under Effect Curve (AUE) From 0-2 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h post-dose
Sleepy: Area Under Effect Curve (AUE) From 0-8 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Dizzy: Area Under Effect Curve (AUE) From 0-1 Hour | pre-dose, 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Dizzy VAS assesses the effect experienced by the participant on a 100-point unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0) to 'extremely' (score of 100).
Dizzy: Area Under Effect Curve (AUE) From 0-2 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h post-dose
Dizzy: Area Under Effect Curve (AUE) From 0-8 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Any Drug Effects: Peak Effect (Emax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Good Drug Effects: Peak Effect (Emax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Bad Drug Effects: Peak Effect (Emax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Feel Sick: Peak Effect (Emax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Nausea: Peak Effect (Emax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Sleepy: Peak Effect (Emax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Dizzy: Peak Effect (Emax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Pupillometry: Area Under Effect Curve (AUE) From 0-1 Hour | pre-dose, 5 min, 15 min, 30 min, 45 min, 1 h post-dose
  Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants have the size of their pupil measured (in mm) using a pupillometer. Measurements are made in a dimly lit (mesopic) room with controlled lighting conditions.
Pupillometry: Area Under Effect Curve (AUE) From 0-2 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2 h post-dose
Pupillometry: Area Under Effect Curve (AUE) From 0-8 Hours | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8 h post-dose
Pupillometry: Peak Effect (Emax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Pupillometry: Time to Maximum (Peak) Effect (TEmax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Drug Liking: Time to Maximum (Peak) Effect (TEmax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
High: Time to Maximum (Peak) Effect (TEmax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Any Drug Effects: Time to Maximum (Peak) Effect (TEmax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Good Drug Effects: Time to Maximum (Peak) Effect (TEmax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Bad Drug Effects: Time to Maximum (Peak) Effect (TEmax) | 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Sleepy: Time to Maximum (Peak) Effect (TEmax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Dizzy: Time to Maximum (Peak) Effect (TEmax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Nausea: Time to Maximum (Peak) Effect (TEmax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Feel Sick: Time to Maximum (Peak) Effect (TEmax) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Plasma Concentration of Oxycodone 5 Minutes Post-Dose (C5min) | pre-dose, 5 min post-dose
Plasma Concentration of Oxymorphone 5 Minutes Post-Dose (C5min) | pre-dose, 5 min post-dose
Plasma Concentration of Noroxycodone 5 Minutes Post-Dose (C5min) | pre-dose, 5 min post-dose
Plasma Concentration of Naltrexone 5 Minutes Post-Dose (C5min) | pre-dose, 5 min post-dose
Plasma Concentration of 6-beta-naltrexol 5 Minutes Post-Dose (C5min) | pre-dose, 5 min post-dose
Plasma Decay Half-Life (t1/2) of Oxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Plasma Decay Half-Life (t1/2) of Oxymorphone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Plasma Decay Half-Life (t1/2) of Noroxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Plasma Decay Half-Life (t1/2) of Naltrexone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Plasma Decay Half-Life (t1/2) of 6-beta-naltrexol | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Oxycodone Concentration-Time Curve (AUC0-1h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
  AUC is a measure of the plasma concentration of the drug over time.
Area Under the Oxymorphone Concentration-Time Curve (AUC0-1h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Noroxycodone Concentration-Time Curve (AUC0-1h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Naltrexone Concentration-Time Curve (AUC0-1h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the 6-beta-naltrexol Concentration-Time Curve (AUC0-1h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Oxycodone Concentration-Time Curve (AUC0-2h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Oxymorphone Concentration-Time Curve (AUC0-2h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Noroxycodone Concentration-Time Curve (AUC0-2h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Naltrexone Concentration-Time Curve (AUC0-2h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the 6-beta-naltrexol Concentration-Time Curve (AUC0-2h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Oxycodone Concentration-Time Curve (AUC0-8h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Oxymorphone Concentration-Time Curve (AUC0-8h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Noroxycodone Concentration-Time Curve (AUC0-8h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Naltrexone Concentration-Time Curve (AUC0-8h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the 6-beta-naltrexol Concentration-Time Curve (AUC0-8h) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero to Last Quantifiable Oxycodone Concentration (AUClast) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero to Last Quantifiable Oxymorphone Concentration (AUClast) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero to Last Quantifiable Noroxycodone Concentration (AUClast) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero to Last Quantifiable Naltrexone Concentration (AUClast) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero to Last Quantifiable 6-beta-naltrexol Concentration (AUClast) | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero Extrapolated to Infinity (AUCinf) for Oxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero Extrapolated to Infinity (AUCinf) for Oxymorphone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero Extrapolated to Infinity (AUCinf) for Noroxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero Extrapolated to Infinity (AUCinf) for Naltrexone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Area Under the Curve From Time Zero Extrapolated to Infinity (AUCinf) for 6-beta-naltrexol | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Systemic Clearance (Cl) of Oxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Systemic Clearance (Cl) of Oxymorphone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Systemic Clearance (Cl) of Noroxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Systemic Clearance (Cl) of Naltrexone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Systemic Clearance (Cl) of 6-beta-naltrexol | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Volume of Distribution at Steady State (Vss) for Oxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Volume of Distribution at Steady State (Vss) for Oxymorphone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Volume of Distribution at Steady State (Vss) for Noroxycodone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Volume of Distribution at Steady State (Vss) for Naltrexone | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Volume of Distribution at Steady State (Vss) for 6-beta-naltrexol | pre-dose, 5 min, 15 min, 30 min, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Salt Lake City, Utah, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4981002&StudyName=A%20Study%20to%20Characterize%20the%20Abuse%20Liability%20of%20Intravenous%20Oxycodone%20Alone%20or%20in%20Combination%20with%20Intravenous%20Naltrexone%20in%20Healthy%2C%20N